CLINICAL TRIAL: NCT02853487
Title: Circadian Rhythm and Attack-timing in Episodic Cluster Headache Patients in- and Outside of Bout: an Actigraphic Study
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, MD, Ph.d.-student Nunu Lund, MD, PhD-student, Danish Headache Center
Other Study IDs: H-7-2014-020
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Cluster Headache
Keywords: Cluster headache; actigraphy; circadian rhythm
MeSH Terms: conditions — Cluster Headache | interventions — Actigraphy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cluster headache patients: Episodic cluster headache patients in- and outside of bout will wear an actigraph and fill out a diary for 2 weeks.
  Interventions: Device: Actigraphy; Other: Diary
- Control group: Healthy, headache-free controls will wear an actigraph and fill out a diary for 2 weeks.
  Interventions: Device: Actigraphy; Other: Diary

INTERVENTIONS:
Device: Actigraphy — An actigraph from Philips
  Other Names: Actigraph from Philips
Other: Diary — Questions on sleep times and awakenings and attacks in the morning and evening for 2 weeks.

SUMMARY:
The aim is to investigate circadian rhythm in episodic cluster headache using actigraphy.

DETAILED DESCRIPTION:
The aim is to investigate circadian rhythm in episodic cluster headache patients in- and outside of bout. This will be done using actigraphy and a short diary for 2 weeks in each period. A secondary outcome is to look at attack occurence and physical activity before and during an attack.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Age between 18 and 65 years of age
* Episodic cluster headache
* The patient can differentiate cluster headache from other primary headaches if he suffers from any.

Exclusion Criteria:

* Circumstances, determined by the PI, that makes the patient ineligible.
* Changes in preventive medication within 7 days before the study initiation and during the 2 weeks.
* Changes in antidepressive medication or antipsychotic medication within 2 weeks before the study initiation and during the 2 weeks.
* Serious somatic and/or psychiatric disorders
* Alcohol intake > 50 units pr.week
* Pregnancy / breastfeeding
* Patient cannot accept the conditions of the trial
* Patient does not understand Danish.

CONTROLS

Inclusion Criteria:

- Age between 18 and 65 years of age

Exclusion Criteria:

* Circumstances, determined by the PI, that makes the patient ineligible.
* Any primary headache more than 1 day / month
* Diagnosed with a secondary headache
* Treatment with antidepressive medication or antipsychotic medication within 2 weeks before the study initiation and during the 2 weeks.
* Serious somatic and/or psychiatric disorders
* Alcohol intake > 14 / 7 units pr.week (males / females)
* Pregnancy / breastfeeding
* Patient cannot accept the conditions of the trial
* Patient does not understand Danish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with episodic cluster headache as defined by ICHD III beta
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Circadian rhythm | Circadian rhythm is assessed after 2 weeks
  After 2 weeks of actigraphy, the circadian rhythm will be assessed using "Philips Actiware 6" program.

SECONDARY OUTCOMES:
Attack occurence | The time of day will be assessed after 2 weeks
Physical activity before and during an attack | Increase / decrease in activity count will be described after 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Rigmor Jensen, Professor, Principal Investigator — Danish Headache Centerq
Locations (1):
- Danish Headache Center, Dept. of Neurology, Rigshospitalet -Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lund NL, Snoer AH, Jennum PJ, Jensen RH, Barloese MCJ. Sleep in cluster headache revisited: Results from a controlled actigraphic study. Cephalalgia. 2019 May;39(6):742-749. doi: 10.1177/0333102418815506. Epub 2018 Nov 23. PMID 30470143